CLINICAL TRIAL: NCT06995066
Title: A Study on the Treatment of Cervical Disc Herniation by Low-temperature Plasma Radiofrequency Ablation Combined With Ozone Injection and Collagenase
Brief Title: Combined Therapy for Cervical Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchong Central Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NanchongCH
Record Dates: First submitted 2025-05-10; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: VAS and JOA Scores; Adverse Reaction Rates; Clinical Efficacy at 1 Month and 6 Months

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): The study group received low-temperature plasma radiofrequency ablation and ozone injection as the control group, with the addition of collagenase injection into the epidural space.
  Interventions: Procedure: collagenase injection into the epidural space
- Control Group (Experimental): The control group underwent low-temperature plasma radiofrequency ablation combined with ozone injection.
  Interventions: Procedure: collagenase injection into the epidural space

INTERVENTIONS:
Procedure: collagenase injection into the epidural space — The "Collagenase injection into the epidural space" is a medical procedure for treating cervical disc herniation. Firstly, the patient is positioned, and the specific location of the epidural space at the affected cervical spine segment is accurately identified with the guidance of imaging devices like fluoroscopy or CT. After local anesthesia, a special puncture needle is inserted into the epidural space following the marked path. Once the needle is in the correct position, an appropriate amount of collagenase solution is slowly injected. After the operation, the patient needs to stay in the hospital for observation to monitor vital signs and neurological conditions. The patient should rest in bed for a certain period and then gradually engage in proper activities. Additionally, personalized rehabilitation treatment plans, including physical therapy and exercise, are usually required to help with recovery.

SUMMARY:
This study mainly explores the efficacy and safety of low-temperature plasma radiofrequency ablation combined with ozone injection and collagenase in the treatment of cervical disc herniation.The primary outcomes included the collection of clinical data for all patients, such as gender, age, surgical segment, preoperative scores, and VAS and JOA scores at 1 week, 1 month, 3 months, and 6 months postoperatively, as well as a comparison of adverse reaction rates between the two groups. The secondary outcomes involved evaluating clinical efficacy at 1 month and 6 months after surgery using the modified Macnab criteria.

DETAILED DESCRIPTION:
1. Research Objective This study mainly explores the efficacy and safety of low-temperature plasma radiofrequency ablation combined with ozone injection and collagenase in the treatment of cervical disc herniation. By establishing this objective, the study sets the overall direction, aiming to comprehensively evaluate how this combined treatment impacts the therapeutic outcomes and safety profile of patients suffering from cervical disc herniation. This objective serves as the cornerstone, guiding the selection of outcome measures, data collection methods, and the overall research design.
2. Primary Outcome Measures The primary outcomes included the collection of clinical data for all patients, such as gender, age, surgical segment, preoperative scores, and VAS and JOA scores at 1 week, 1 month, 3 months, and 6 months postoperatively, as well as a comparison of adverse reaction rates between the two groups. Firstly, the collection of comprehensive clinical data from all participants, including demographic information like gender, age, and the specific surgical segment, provides a detailed characterization of the patient cohort. This baseline data is crucial for understanding the patient population's characteristics, enabling researchers to account for potential confounding factors during data analysis and ensuring the validity of the study results.

   Secondly, the collection of preoperative scores, along with Visual Analog Scale (VAS) and Japanese Orthopaedic Association (JOA) scores at multiple postoperative time points (1 week, 1 month, 3 months, and 6 months), allows for a dynamic assessment of treatment efficacy. The VAS scores track the evolution of pain levels over time, offering a direct measure of how effectively the treatment alleviates patients' discomfort. Meanwhile, the JOA scores evaluate the recovery of cervical spine function, providing insights into the overall improvement of patients' quality of life and functional ability. By monitoring these scores at different intervals, researchers can observe the treatment's short-term and long-term effects, identify trends in patient recovery, and determine the optimal time frame for achieving the best outcomes.

   Lastly, the comparison of adverse reaction rates between the two groups is a pivotal component for evaluating treatment safety. By systematically documenting and contrasting the occurrence of adverse events, such as allergic reactions, infections, or neurological complications, researchers can determine whether the combined treatment poses a higher risk to patients. This comparison helps in balancing the potential benefits of the treatment against its associated risks, guiding clinical decision-making and ensuring patient well-being.
3. Secondary Outcome Measures The secondary outcomes involved evaluating clinical efficacy at 1 month and 6 months after surgery using the modified Macnab criteria. Utilizing the modified Macnab criteria to evaluate clinical efficacy at 1 month and 6 months post-surgery provides a standardized, comprehensive framework for gauging treatment success. This criteria assesses multiple dimensions of patient recovery, including symptom relief, functional improvement, and patient satisfaction. By incorporating a broader range of factors beyond just pain and function scores, it offers a more holistic understanding of the treatment's impact on patients' overall condition. This secondary evaluation complements the primary outcome measures, providing additional evidence to support the study's findings and enhancing the robustness of the conclusions regarding the combined treatment's efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with cervical disc herniation through MRI or CT, with single-level disc protrusion (C3-C7) that occupies ≤1/3 of the central spinal canal.
* Aged between 30 and 80 years.
* Have suffered from persistent neck/shoulder pain or upper extremity radiating pain for ≥3 months.
* The pain does not respond to conventional treatments, including traction, massage, and oral medications.
* Be willing to undergo surgery therapy.
* Have no prior cervical spine surgery.

Exclusion Criteria:

* Cervical instability, myelopathic spondylosis, severe spinal stenosis (canal occupancy >1/3), or ligament calcification.
* Severe osteoporosis (T-score <-2.5).
* Extruded or sequestered disc herniation
* Coagulation disorders or active infections
* Cervical deformities, tumors, or a history of cervical spine surgery

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) score at 1 week, 1 month, 3 months, and 6 months postoperatively, as well as a comparison of adverse reaction rates between the two groups. | 6 months
  The Visual Analogue Scale (VAS) score is a psychometric tool used to measure subjective experiences such as pain, anxiety, or satisfaction.
  The following is a detailed description of the meanings represented by specific numerical values in the VAS score, typically converted to a 0-10 numerical scale for clinical use:
  0: Represents the complete absence of the measured sensation (e.g., pain) 1-2: Very mild level. Sensation is barely noticeable and does not interfere with daily activities.
  3: Mild but distinct sensation. Noticeable enough to be recognized but still easily ignored or managed.
  Moderate level. 4-6: Moderate level. Sensation is clearly present and affects daily activities to some extent, but remains tolerable.
  7-9: Severe level. Sensation dominates attention and drastically limits functionality; immediate intervention may be needed.
  10: Maximal/intolerable level. Sensation is beyond endurance, rendering the individual unable to perform any normal activities.

SECONDARY OUTCOMES:
evaluating clinical efficacy at 1 month and 6 months after surgery using the modified Macnab criteria | 6 months
  The modified Macnab criteria is a clinical scoring system used to evaluate the outcome of spinal surgeries by assessing patient satisfaction, symptom relief, and functional status. Below is a description of the specific numerical values and their meanings, typically categorized into excellent, good, fair, and poor outcomes:
  Excellent: Symptoms: Complete resolution of pain and neurological deficits (e.g., weakness, numbness).
  Good: Symptoms: Significant improvement in pain and neurological symptoms, with only mild residual issues.
  Fair: Symptoms: Moderate improvement, but persistent pain or neurological deficits that affect quality of life.
  Poor: Symptoms: Little to no improvement, or symptoms may have worsened post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanchong Central Hospital, Nanchong, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
Ethical and Legal Constraints Informed Consent Limitations: Participants in prospective studies have not explicitly consented to broader data sharing.
  Ethical Risks: Even with de-identification, residual identifiability risks (e.g., through rare demographic or clinical data) may raise ethical concerns about re-identification of participants.